CLINICAL TRIAL: NCT02598648
Title: Daping Hospital of the Third Military Medical University
Brief Title: Role and Molecular Mechanism of Farnesoid X Receptor(FXR) and RIPK3 in the Formation of Acute Respiratory Distress Syndrome in Neonates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Fang Wu, Principal Investigator Fang Wu, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 8157060555
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Lung Injury; FXR; RIPK3
Keywords: FXR; RIPK3; Neonates; Acute Respiratory Distress Syndrome; Acute Lung Injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ALI( acute lung injury) (Other): Diagnostic criteria: 1.Acute onset；2.FiO2/ PaO2< 40.0 kPa (300mmHg, ALI); 3.Chest X-ray showed that the double lung texture increased, the increase of crude, fuzzy, visible diffuse patchy infiltration shadow with compensatory emphysema, for the most early performance; B. double lung field large sheet, asymmetric, edge fuzzy infiltration shadow, the most dense in the lung；4. Echocardiography, left atrial hypertension; 5.The gestational age >35 week, have maternal age cholestasis (severe), sepsis or meconium aspiration syndrome (MAS) understanding of history, and with the exception of the primary pulmonary surfactant (PS) lack of. FXR and RIPK3 were measured in neonate with ALI.
  Interventions: Other: FXR; Other: RIPK3
- ARDS(respiratory distress syndrome) (Other): ARDS :Diagnostic criteria: 1.Acute onset；2.FiO2/ PaO2< 26.7 kPa (200mmHg, ARDS); 3.Chest X-ray showed that the double lung transparent brightness is generally lower, the glass sample, with bronchial inflatable sign, and even double lung field common density increased, the heart shadow is not clear, a white lung, as the most important performance；4. Echocardiography, left atrial hypertension; 5.The gestational age >35 week, have maternal age cholestasis (severe), sepsis or meconium aspiration syndrome (MAS) understanding of history, and with the exception of the primary pulmonary surfactant (PS) lack of；6.Need to use a ventilator.
  FXR and RIPK3 were measured in neonate with ALI.were measured in another group neonate with ARDS
  Interventions: Other: FXR; Other: RIPK3
- control (Other): Control group: Patients with mechanical ventilation due to external causes of the lung, no ALI-ARDS performance,FiO2/ PaO2< 40.0 kPa (300 mmHg), such as premature apnea or HIE. FXR and RIPK3 were measured in neonate with HIE
  Interventions: Other: FXR; Other: RIPK3

INTERVENTIONS:
Other: FXR — FXR could elevate the transcription of RIPK3, a key protein in necroptosis, and play important role in bile aicd induced alveolar epithelial cell(AEC) necroptosis. FXR were measured in neonate with ALI、ARDS and control
Other: RIPK3 — FXR(farnesoid-X-receptor) could elevate the transcription of RIPK3, a key protein in necroptosis, and play important role in bile aicd induced alveolar epithelial cell(AEC) necroptosis. RIPK3 were measured in neonate with ALI、ARDS and control.

SUMMARY:
In the clinical data, the changes of RIPK3 and FXR were monitored in the lung lavage fluid and blood from the patients.

In vivo experiments to find high risk factors to induce AEC necrosis and further lead to ARDS evidence, can provide a more direct theoretical research foundation for the pathogenesis of ARDS.

DETAILED DESCRIPTION:
Divided into 3 Arms ALI :Diagnostic criteria: 1.Acute onset；2.FiO2/ PaO2< 40.0 kPa (300mmHg, ALI); 3.Chest X-ray showed that the double lung texture increased, the increase of crude, fuzzy, visible diffuse patchy infiltration shadow with compensatory emphysema, for the most early performance; B. double lung field large sheet, asymmetric, edge fuzzy infiltration shadow, the most dense in the lung；4. Echocardiography, left atrial hypertension; 5.The gestational age >35 week, have maternal age cholestasis (severe), sepsis or meconium aspiration syndrome (MAS) understanding of history, and with the exception of the primary pulmonary surfactant (PS) lack of.

ARDS :Pediatric acute respiratory distress syndrome (ARDS) is a severe lung injury caused by pneumonia, sepsis, and trauma.Diagnostic criteria: 1.Acute onset；2.FiO2/ PaO2< 26.7 kPa (200mmHg, ARDS); 3.Chest X-ray showed that the double lung transparent brightness is generally lower, the glass sample, with bronchial inflatable sign, and even double lung field common density increased, the heart shadow is not clear, a white lung, as the most important performance；4. Echocardiography, left atrial hypertension; 5.The gestational age >35 week, have maternal age cholestasis (severe), sepsis or meconium aspiration syndrome (MAS) understanding of history, and with the exception of the primary pulmonary surfactant (PS) lack of；6.Need to use a ventilator.

Control group: Patients with mechanical ventilation due to external causes of the lung, no ALI-ARDS performance,FiO2/ PaO2< 40.0 kPa (300 mmHg), such as premature apnea or HIE.

ELIGIBILITY:
Inclusion Criteria:According to the diagnostic criteria, the diagnosis was ALI or ARDS； Exclusion Criteria:Severe congenital or hereditary disease of the newborn, is clearly diagnosed as NRDS, which is caused by the lack of the primary PS。

Max Age: 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2015-09-20; Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
FXR | 6 hours later

SECONDARY OUTCOMES:
chest-X-ray | 1 hours later
RIPK3 | 6 hours later
blood gas | 1 hours later

CONTACTS AND LOCATIONS:
Overall Officials: Hu Zh Xue, Doctorate, Study Director — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- NICU of Daping Hospital of the Third Military Medical University, Chongqing, Chongqing Municipality, China